CLINICAL TRIAL: NCT06603090
Title: Text4Vax: Understanding the Effectiveness and Implementation of Text Message Reminders for Pediatric COVID-19 and Influenza Vaccines 2024-2025 Season
Brief Title: Text4Vax: Text Message Reminders for Pediatric COVID-19 and Influenza Vaccines 2024-25 Season
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Children's Hospital of Philadelphia (Other); American Academy of Pediatrics (Other); University of Pennsylvania (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Melissa Stockwell, Professor of Pediatrics; Professor of Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: AAAV0563-01; 1R01AI182165 (NIH)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Influenza; COVID-19; Vaccination Hesitancy
Keywords: text message; Short message service (SMS); mHealth
MeSH Terms: conditions — Influenza, Human; COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Text message influenza and COVID-19 vaccine reminders (Experimental): Text message reminders for both influenza and COVID-19 vaccinations
  Interventions: Behavioral: Text message influenza and COVID-19 vaccine reminders
- Text message influenza vaccine reminders (Experimental): Text message reminders only for influenza vaccination
  Interventions: Behavioral: Text message influenza vaccine reminders
- Text message COVID-19 vaccine reminders (Experimental): Text message reminders only for COVID-19 vaccination
  Interventions: Behavioral: Text message COVID-19 vaccine reminders
- Usual Care (No Intervention): Usual care has no text message

INTERVENTIONS:
Behavioral: Text message influenza vaccine reminders — Text message influenza vaccine reminders
  Arms: Text message influenza vaccine reminders
Behavioral: Text message COVID-19 vaccine reminders — Text message COVID-19 vaccine reminders
  Arms: Text message COVID-19 vaccine reminders
Behavioral: Text message influenza and COVID-19 vaccine reminders — Text message influenza and COVID-19 vaccine reminders
  Arms: Text message influenza and COVID-19 vaccine reminders

SUMMARY:
This multi-site study assesses the impact of text message reminders on the receipt of COVID-19 and influenza text message reminders takes place primarily in practices from the American Academy of Pediatrics (AAP) Pediatric Research in Office Settings (PROS) network.

DETAILED DESCRIPTION:
The study is to be conducted over the 1st season (September 2024-April 2025) as an effectiveness trial and the 2nd (September 2025-April 2026) as a replication study. This protocol covers the first season. Parents of eligible children who are 6 month-17 year-old who are due for both a COVID-19 and influenza vaccine will be sent text messages. Within each practice site, parents of eligible children will be randomized to receive either: 1) combined COVID-19 and influenza vaccine text message reminders, 2) COVID-19 reminders alone, 3) influenza reminders alone, or 4) no reminders (usual care).

Randomization is to be stratified by practice site, age group and prior year's COVID-19/influenza vaccine history. Messages will be sent centrally and managed by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Child that:

  * is 6 months-17 year-old children
  * due for both a COVID-19 and influenza vaccine
* Receives care at study site
* Language listed in electronic health record is English or Spanish
* Has not opted out of text messages from practice

Exclusion Criteria:

* Has opted out of text messages from practice
* Language listed in electronic health record is not English or Spanish

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66147 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Timeliness of influenza vaccination | Up to December 31 each year, up to ~90 days
  Days from study start to influenza vaccine up to December 31 each year
Timeliness of COVID-19 vaccination | Up to December 31 each year, up to ~90 days
  Days from study start to COVID-19 vaccine up to December 31 each year

SECONDARY OUTCOMES:
Timeliness of influenza vaccination | Up to April 30 each year, up to ~210 days
  Days from study start to influenza vaccine up to April 30 each year
Timeliness of COVID-19 vaccination | Up to April 30 each year, up to ~210 days
  Days from study start to COVID-19 vaccine up to April 30 each year
Percentage of Participants Who Received Influenza Vaccine by December 31 Each Year | ~3 months
  Receipt of influenza vaccine by December 31 each year
Percentage of Participants Who Received COVID-19 Vaccine by December 31 Each Year | ~3 months
  Receipt of COVID-19 vaccine by December 31 each year
Percentage of Participants Who Received Influenza Vaccine by April 30 Each Year | ~7 months
  Receipt of influenza vaccine by April 30 each year
Percentage of Participants Who Received COVID-19 Vaccine by April 30 Each Year | ~7 months
  Receipt of COVID-19 vaccine by April 30 each year

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University; Alex Fiks, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - American Academy of Pediatrics, Itasca, Illinois
  - Columbia University Irving Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No